CLINICAL TRIAL: NCT00495313
Title: Determine the Effects of COL-101 Administered Once Daily With Metronidazole Topical Gel, 1% Versus Doxycycline Hyclate 100 mg Administered Once Daily With Metronidazole Topical Gel, 1% in Patients With Moderate to Severe Rosacea
Brief Title: Safety and Efficacy Study to Compare Two Rosacea Treatment Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CollaGenex Pharmaceuticals (Industry)
Responsible Party: C. Powala, VP, Drug Development & Regulatory Affairs, CollaGenex Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: COL101-ROSE-401
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: doxycycline (Active Comparator): Vibramycin plus metronidazole
  Interventions: Drug: doxycycline
- Cohort 2 (Active Comparator): Oracea® delayed release plus metronidazole
  Interventions: Drug: doxycycline

INTERVENTIONS:
Drug: doxycycline — COL-101, QD plus metronidazole
  Other Names: Vibramycin, 100 mg, QD plus metornidazole
  Arms: Cohort 1: doxycycline
Drug: doxycycline — 40 mg with metronidazole QD
  Other Names: Oracea® 40 mg plus metronidazole
  Arms: Cohort 2

SUMMARY:
To compare the safety and efficacy of two treatment regimens: 1) COL-101 and metronidazole gel 1%; 2) Doxycycline hyclate 100 mg and metronidazole gel 1%

DETAILED DESCRIPTION:
Compare the safety and efficacy of two treatment regimens: 1) COL-101 and metronidazole gel 1%; 2) Doxycycline hyclate 100 mg and metronidazole gel 1%

ELIGIBILITY:
Inclusion Criteria:

* 8-40 total lesions
* erythema
* telangiectasia

Exclusion Criteria:

* non-pregnant, non-lactating
* achlorhydric
* gastric by-pass surgery
* allergy to study medications
* drug/alcohol abuse
* use of proton pump inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in total lesion count from Baseline at the study endpoint | 16 weeks

SECONDARY OUTCOMES:
Change in Investigator's Global Assessment from Baseline at the study endpoint | 16 weeks
Change in Clinician's Erythema Assessment score from Baseline at the study endpoint | 16 weeks
Change in total lesion count (papules + pustules + nodules) from Baseline at each visit | 4 weeks, 8 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Powala, JD, Study Chair — CollaGenex Pharmaceuticals
Locations (7):
- United States (7):
  - Joel Schlessinger, Omaha, Nebraska
  - James Del Rosso, Las Vegas, Nevada
  - Angela Moore, Arlington, Texas
  - William Abramovits, Dallas, Texas
  - Douglas Forsha, West Jordan, Utah
  - Bernard Goffe, Seattle, Washington
  - William Werschler, Spokane, Washington